CLINICAL TRIAL: NCT04658030
Title: 360° Video VR Surgery Preparation: Feasibility, Acceptability, Tolerability and Initial Effectiveness of Virtual Reality for Children in a Flemish Hospital.
Brief Title: Immersive Care - Virtual Reality(VR) 360 Pediatric Surgery Preparation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas More University of Applied Sciences (Other)
Collaborators: Heilig Hart Ziekenhuis Lier (Unknown); Fotosfeer (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IC_PED_2
Record Dates: First submitted 2020-11-09; First posted 2020-12-08 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Surgery
Keywords: Pediatrics; Preparation; Virtual Reality; 360 Video; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR 360 video surgery preparation (Experimental): Preparing pediatric patients for surgery with a newly developed VR 360 degree video. Maximum 30 minutes, one time.
  Interventions: Device: VR 360 video surgery preparation
- Care as usual (Active Comparator): Preparing the children for surgery with the care as usual. A booklet that can be viewed by the children and parents at home.
  Interventions: Other: Care as usual

INTERVENTIONS:
Device: VR 360 video surgery preparation — Preparing children on the surgery by a virtual reality 360 degrees video tour from the pediatric ward to the surgery room. In this video all information is given necessary for the surgery. This takes a maximum of 30 minutes and will be performed 1 time.
  Arms: VR 360 video surgery preparation
Other: Care as usual — Preparing the children for surgery with the care as usual. A booklet that can be viewed by the children and parents at home.
  Arms: Care as usual

SUMMARY:
Context: This study is part of the larger Immersive Care project which (in short) seeks the connection between technology and care by conducting feasibility studies with promising technological interventions tailored to care.

This is one of the case studies from the larger project titled: 360 ° video VR surgery preparation: feasibility, acceptability, tolerability and initial effectiveness of virtual reality for children in a Flemish hospital.

Domain: This scientific study will take place in 1 hospital on the pediatric ward. The target group consists of children between 6 and 12 years of age who will undergo an operation, the parents and the care providers involved.

Target:

1. Assess the acceptability, feasibility and tolerability of the 360 ° video VR surgery preparation.
2. Assess the effectiveness of the 360 ° video VR surgery preparation on preoperative procedural anxiety in children, comparing the intervention with care as usual (CAU *).

   * CAU in this study is a picture book which is a kind of animated video with text to explain what will happen on the day of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained
* Inpatient or outpatient in the study site (Heilig Hart Hospital Lier): each paediatric patient who will undergo surgery during the study period (01-12-2020 and 30-09- 2021).
* Age range of ≥ 6 and ≤ 12
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing

Exclusion Criteria:

* Patient has a history of seizure disorders (e.g. epilepsy)
* Physical impairment that preclude VR intervention (e.g. facial burns or wounds, contagious infectious disease, need for intensive care)
* Non-Dutch/English/French speaker: Both the paediatric patient and his/her caregiver must be able to provide informed consent and assent
* Previous enrolment in this study (during a previous hospital stay)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in staff attitude towards the intervention | Staff: Measurement takes place in week 5 after the start of the study.
  Unified theory of acceptance and use of technology tests the acceptance of the staff towards the intervention in this study.
  Assess change in patient attitude towards the intervention with the Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire survey. The UTAUT questionnaire survey for end-users consists of 20 items with five response options ranging from "Totally disagree" to "Totally agree". The questionnaire survey consists of 7 subscales, for most of which higher scores indicate a more positive attitude towards the intervention.
Change from baseline in tolerability (Do participants experience symptoms of simulator sickness?) | Immediately after the intervention
  Assessment of physical side effects after exposure to VR by the Pediatric Simulator Sickness Questionnaire (Peds SSQ).
  The Peds SSQ contains queries that probe 4 symptom categories: (1) eye strain (queries 1-4); (2) head and neck discomfort (queries 5 and 6); (3) sleepiness (solipsism) or fatigue (queries 7 and 8); and dizziness or nausea (visually induced motion sickness, queries 9-13). The scale that is used is a likert scale (with additional faces) ranging from 0 to 6 per query (0 = no of the above "complaints"; 6 = a lot of the above "complaints".
Usability of the intervention: System Usability Scale (SUS) | Immediately after the intervention.
  Assessment of ease of use of the intervention with the System Usability Scale (SUS). The SUS is a 10 item questionnaire with five response options for respondents; from "strongly disagree" to "strongly agree". A higher SUS score indicates better usability.
Patient satisfaction: Client Satisfaction Questionnaire (CSQ-8) | Immediately after the intervention
  Assessment of client satisfaction with the VR application with the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 consists of 8 items with four response options. Higher scores indicate higher satisfaction.
Intervention adherence | Immediately after the intervention
  Measure intervention adherence by registering the number of fully completed sessions.
Procedure time | Immediately after the intervention
  The procedure time of intervention in minutes

SECONDARY OUTCOMES:
Preliminary effectiveness (change in anxiety between timepoints) (Intervention and control) | Measurement 1: Immediately after signing the informed consent, day 1 of study. Measurement 2: Immediately after the intervention, day 1 of study. Measurement 3: Just before surgery, day 4 of study
  Measuring procedural anxiety (with a Visual Analogue Scale) (1.Before intervention/control, 2. just after intervention/control and 3.just before surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Wessel van de Veerdonk, PhD, Principal Investigator — Thomas More University of Applied Sciences
Locations (1):
- Heilig Hart Ziekenhuis Lier, Lier, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No